CLINICAL TRIAL: NCT04736654
Title: Cross-cultural Adaptation, Reliability and Validity of the Turkish Version of the Headache Disability Questionnaire
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Halime ARIKAN, Research Assistant, Gazi University
Other Study IDs: 83116987-569
Record Dates: First submitted 2021-01-30; First posted 2021-02-03 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2023-09

CONDITIONS: Headache; Headache Disorders; Headache, Migraine; Headache, Tension; Headaches Chronic; Headaches Muscular
Keywords: Headache; Reliability; Validity; Cross-cultural adaptation
MeSH Terms: conditions — Headache; Headache Disorders; Migraine Disorders; Tension-Type Headache | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients group: Individuals with headache
  Interventions: Other: Survey study

INTERVENTIONS:
Other: Survey study — Headache Disability Questionnaire (HDQ) will be applied.

SUMMARY:
The purpose of this study was to investigate cultural adaptation, reliability and validity of the Turkish version of the Headache Disability Questionnaire (HDQ).

DETAILED DESCRIPTION:
When the outcome criteria for the physiotherapy of headache are considered in clinical studies and practice, parameters such as headache frequency, duration and severity are frequently used. Physiotherapists treat musculoskeletal dysfunction in various types of headache, including migraine, tension headache, and cervicogenic headache. The Headache Disability Questionnaire (HDQ), which was developed to measure the quality of life of a general population receiving physiotherapy and experiencing headache, evaluates the pain intensity, daily life activities, disruptions in work or school life, and the influence of the recreational activities of individuals. HDQ consists of 9 items and each item is rated between 0 and 10. Increasing the score indicates the seriousness of the impact. The study is planned with 45 individuals with gluteal tendinopathy. After questioning the sociodemographic characteristics of the individuals, the patients will be asked to fill in HDQ, Migraine Disability Assessment Questionnaire, Headache Impact Test-6 and Short Form-36.Test-retest will be re-applied to those of the same individuals who can be reached after 1 week. The results will be analyzed using the SPSS version 22.0 computer package program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with any type of headache,
* Have a chronic headache.

Exclusion Criteria:

* Having a cognitive and neurological disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals with any type of headache.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Headache Disability Questionnaire (HDQ) | 10 minutes
  Headache Disability Questionnaire is designed to measure the quality of life related to the disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Halime ARIKAN, Ankara, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Derived] Arikan H. Headache Disability Questionnaire: cross-cultural adaptation and validation of the Turkish version. BMC Neurol. 2024 Dec 18;24(1):480. doi: 10.1186/s12883-024-03987-4. PMID 39696036